CLINICAL TRIAL: NCT00640497
Title: A Phase I/II Multicentric Study to Determine the Safety and Efficacy of a Combination of Anti-CD3 & Anti-CD7 Ricin A Immunotoxins for the Treatment of Steroid-Resistant Acute Graft-Versus-Host Disease
Brief Title: Anti-CD3 & Anti-CD7 Ricin A Immunotoxin-Combination for Acute Graft Versus Host Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unavailability of investigational product
Sponsor: Henogen (Industry)
Responsible Party: Sophie Houard CSO, Henogen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN019/ITC-001
Record Dates: First submitted 2008-03-04; First posted 2008-03-21 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Acute Graft Versus Host Disease
Keywords: acute GVHD; immunotoxin; anti-CD3; anti-CD7; Ricin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Treatment arm
  Interventions: Biological: IT-Combination

INTERVENTIONS:
Biological: IT-Combination — The treatment consists of a standard dose of 4 infusions of IT-combination (4 mg/m2), given 48-hours apart over a 4-hour period. The IT-combination is a combination of two immunotoxins. One immunotoxin is a mAb anti-CD3 conjugated to recombinant ricin A chain and the other immunotoxin is a mAb anti-CD7 conjugated to recombinant ricin A chain.

SUMMARY:
In this study, a combination of two T-cell directed antibodies both conjugated to a cell-killing toxin will be evaluated. Previous in vitro studies have demonstrated that this so-called immunotoxin-combination (IT-combination) acts synergistically in eliminating T cells. In a subsequent clinical pilot-study, the IT-combination has generated encouraging results when applied as third line therapy. Extensive biological and clinical responses could be noted in the absence of severe acute toxicities. Building on this experience, the current study aims at evaluating the characteristics of the IT-combination when administered in an earlier phase of the disease, i.e. as second line instead of as third line therapy.

DETAILED DESCRIPTION:
"The experimental design is a non-controlled multicentric fixed-dose Phase I/II study. A total of 12 evaluable patients will be enrolled in 4 transplant centers throughout the Netherlands, in a 9 to 12 months period. The treatment consists of a standard dose of 4 infusions IT-combination (4 mg/m2), given 48-hours apart over a 4-hour period.

The intended follow-up period is 12 months. The patient will also be asked to participate in additional research aiming at determining the presence and evolution of biomarkers suggestive for the extent to which the IT-combination 'resets the T-cell compartment, induces clinical tolerance, and/or enhances the risk of over-immunosuppression."

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from severe acute GVHD (Grade II-IV) progressing after 3 days, or non-improving after 5 days, of prednisolone at 2 mg/kg a day.
* Age ≥ 18 years.
* Patients or their guardians should have given written informed consent using forms approved by the Institutional Review Board.

Exclusion Criteria:

* Patients receiving concomitant investigational therapeutics/prophylaxis for acute GVHD at the time of enrollment.
* Patients with histological signs/symptoms suggestive of chronic GVHD.
* Patients requiring mechanical ventilation, requiring vasopressor support, requiring hemodialysis, having serum creatinine > 266 μmol/l (> 3 mg/dl), or having a serum albumin level of 20 g/l or less.
* Patients having uncontrolled bacterial, viral or fungal infections at the start of therapy.
* Patients with current evidence of active intrapulmonary disease.
* Patients with known hypersensitivity to any of the components of the study drug (murine mAb or RTA).
* Patients who are pregnant, breast feeding, or, if sexually active, unwilling to use effective birth control for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
The acute GVHD response rate on study Day 29 | Day 29

SECONDARY OUTCOMES:
The safety and tolerability of the IT-combination, as determined by the number and intensity of adverse and serious adverse events during 12 months | 12 months
The acute GVHD relapse rate | 12 months
The incidence of chronic GVHD during 12 months | 12 months
The overall survival and progression free survival during 12 months | 12 months
The kinetics of treatment-induced T cell and Natural Killer (NK) cell depletion | 12 months
The pharmacokinetic profile of the IT-combination | day 9
The occurrence and extent of humoral responses against the IT-combination | 12 months
The occurrence of any treatment-induced cytokine release | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Anton V Schattenberg,, MD, PhD,, Principal Investigator — Department of Hematology Radboud University Nijmegen (RUN) Medical Centre
Locations (3):
- Netherlands (3):
  - Department of Hematology Radboud University Nijmegen (RUN), Nijmegen
  - Department of Hematology Erasmus MC/Daniel den Hoed Cancer CenterGroene Hilledijk, Rotterdam
  - L.F. , Department of HematologyUMC Utrecht, Utrecht

REFERENCES:
- [Background] van Oosterhout YV, van Emst L, Schattenberg AV, Tax WJ, Ruiter DJ, Spits H, Nagengast FM, Masereeuw R, Evers S, de Witte T, Preijers FW. A combination of anti-CD3 and anti-CD7 ricin A-immunotoxins for the in vivo treatment of acute graft versus host disease. Blood. 2000 Jun 15;95(12):3693-701. PMID 10845899